CLINICAL TRIAL: NCT02398838
Title: Acceptability and Feasibility of a Simplified Medical Abortion Regimen in Georgia: A Study of 400 mcg Buccal Misoprostol Following 200 mg Mifepristone for Abortion up to 63 Days Gestation
Brief Title: Acceptability and Feasibility of a Simplified Medical Abortion Regimen in Georgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1.2.4.5
Record Dates: First submitted 2014-09-12; First posted 2015-03-26 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Abortion, First Trimester
MeSH Terms: interventions — Mifepristone; Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home administration of mifepristone (Experimental): Home administration of 200 mg mifepristone. Choice of home or clinic administration of 400 mcg buccal misoprostol.
  Interventions: Drug: Home administration of 200 mg mifepristone; Drug: Home or clinic administration of 400 mcg buccal misoprostol
- Clinic administration of mifepristone (Active Comparator): Clinic administration of 200 mg mifepristone. Choice of home or clinic administration of 400 mcg buccal misoprostol.
  Interventions: Drug: Home or clinic administration of 400 mcg buccal misoprostol

INTERVENTIONS:
Drug: Home administration of 200 mg mifepristone — Home administration of 200 mg mifepristone.
  Other Names: Penkrofton
  Arms: Home administration of mifepristone
Drug: Home or clinic administration of 400 mcg buccal misoprostol — Home or clinic administration of 400 mcg buccal misoprostol

SUMMARY:
This study examined the acceptability and feasibility of using a simplified regimen of medical abortion in the eastern and western regions of the country of Georgia. It was hypothesized that home use of mifepristone and buccal administration of misoprostol would be both acceptable and efficacious.

DETAILED DESCRIPTION:
The study recruited women with pregnancies up to 63 days gestation. Eligible women took 200 mg mifepristone. Two days later they took 400 mcg buccal misoprostol, with the option of doing so in the clinic or at home. They underwent clinic follow-up 12-15 days after taking mifepristone to determine if their medical abortions were complete. The study assessed the regimen's efficacy, women's preferences regarding where to administer the medications, and the acceptability of buccal misoprostol and of side effects that accompanied women's medical abortions.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* In good general health
* Living or working close to the study site
* Intrauterine pregnancy less than 64 days gestation
* Willing and able to sign consent forms
* Ready access to a telephone and emergency transportation
* Willing to provide an address and/or telephone number for purposes of follow-up
* Agree to comply with the study procedures and visit schedule

Exclusion Criteria:

* Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass
* IUD in place (IUD must be removed first)
* Chronic renal failure
* Concurrent long-term corticosteroid therapy
* History of allergy to mifepristone, misoprostol or other prostaglandin
* Hemorrhagic disorders or concurrent anticoagulant therapy
* Inherited porphyrias
* Other serious physical or mental health conditions

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 622 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Proportion of abortions that are complete without surgical intervention (unit: percent) | 15 days
  Percentage of women with complete abortion without the need of a surgical intervention.

SECONDARY OUTCOMES:
Proportion of women satisfied with procedure (unit: percent) and with side effects (unit: percent) | 15 days
  Woman's satisfaction with her medical abortion procedure and side effects experienced.

OTHER OUTCOMES:
Proportion of women who select home-use of mifepristone | 1 week
Proportion of women who select home-use of misoprostol | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (4):
- Georgia (4):
  - Batumi Maternity House, Batumi, Adjara
  - Zestafoni Maternity House, Zestaponi, Imereti
  - A. Kambarashvili Clinic, Telavi, Kakheti
  - Bolnisi Maternity House, Bolnisi, Kvemo Kartli